CLINICAL TRIAL: NCT03807258
Title: Functional Implication of Corpus Callosum in Voluntary Strength in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 5 Santé (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5S_PHYCOM
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Neurophysiology; Physiology
Keywords: COPD; Transcranial magnetic stimulation; Motor-evoked potentials; Muscle weakness; Interhemispheric; Inhibition
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness; Inhibition, Psychological | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: COPD Patients vs. Controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD patients group (Experimental): COPD patients undergoing transcranial magnetic stimulation (TMS) evaluations.
  Interventions: Other: Transcranial magnetic stimulation (TMS)
- Controls group (Active Comparator): Healthy matched controls undergoing transcranial magnetic stimulation (TMS) evaluations.
  Interventions: Other: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Other: Transcranial magnetic stimulation (TMS) — Evaluations by TMS

SUMMARY:
Patients with COPD have lower capability of activating their muscles. At the cortical level, force production is not only controlled by contralateral primary motor cortex but also by ipsilateral motor cortex. The aim of this study is to determine whether ipsilateral areas are functionally impaired in COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) patients exhibit not only respiratory symptoms but also a peripheral muscular weakness. This weakness is characterized by a loss in strength, harmful for the patients' life quality and vital prognosis (Swallow et al., 2007). Even if many studies have enlightened damages at a peripheral level, the muscular atrophy itself cannot totally explain the loss in force (Menon et al., 2012). Furthermore, the contractile properties of COPD muscles fibres are preserved (Debigare et al., 2003). Consequently, peripheral muscle weakness cannot only be explained by peripheral factors and central structures must be investigated.

At the central level, it is admitted that force production is controlled by the activation of contralateral motor areas. In COPD, these areas were found to be less activated than in controls during force production (Alexandre et al., 2014). However, recent studies bring the evidence that ipsilateral motor areas are also mobilized to cope demand during such task. The activation of ipsilateral areas is possible through inter hemispheric pathways, as the corpus callosum. Recently, the integrity of the corpus callosum have been linked to the capability of activating the ipsilateral motor cortex (Chiou et al., 2014) during force production. This is of concern knowing that several studies reported white matter lesions in the brain of COPD patients (Dodd et al, 2012) and more precisely in regions containing the corpus callosum (Lahousse et al., 2013).

Therefore, we hypothesize that COPD patients have a lower capability of activating their ipsilateral motor cortex during force production compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Health insurance
* Patients : COPD Gold II-IV

Exclusion Criteria:

* Pregnant women
* Seizures
* Unable to give written consent
* Metalic object above shoulders
* Dermatological issue concerning surface electrodes
* Caffeine consumption > 4 coffee / day
* Neurological disorders
* Opioid-based treatment
* Patients : recent exacerbation (< 4 weeks)
* Patients : rehabilitation in previous 1 year

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Ipsilateral excitability ratio : rest - 50% mvic | Baseline
  Ratio of ipsilateral excitability. Measured at rest, and during a 50% max. isometric contraction. Then, ipsilateral excitability ratio = rest / 50% * 100.

SECONDARY OUTCOMES:
Ipsilateral inhibition ratio : rest - 50% mvic | Baseline
  Ratio of ipsilateral inhibition. Measured at rest, and during a 50% max. isometric contraction. Then, ipsilateral inhibition ratio = rest / 50% * 100. SICI (2ms) method is used to quantify inhibition.
Interhemispheric inhibition | Baseline
  Interhemispheric inhibition, from contralateral to ipsilateral motor cortex, using reference method from Ferbert et al., 1992.
Relationship between inter hemispheric inhibition and voluntary strength | Baseline
  Correlation coefficient between inter hemispheric inhibition and maximal isometric force production
S100B and GFAP | Baseline
  Serum concentrations of S100B and GFAP proteins, brain lesions markers

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Oliver, MD, Principal Investigator — 5 Santé
Locations (2):
- France (2):
  - Cliniques du Souffle, Lodève, Herault
  - Cliniques du Souffle, Osséja, Pyrenees Orientales

IPD SHARING:
Plan to Share IPD: No